CLINICAL TRIAL: NCT04577755
Title: A Multicenter Phase II Study of Pomalidomide Monotherapy in Kaposi Sarcoma
Brief Title: Pomalidomide Treatment in Patients With Kaposi Sarcoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-07565; NCI-2020-07565 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-108 (Other: AIDS Malignancy Consortium); AMC-108 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Skin Kaposi Sarcoma
MeSH Terms: interventions — Biopsy; Specimen Handling; pomalidomide; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pomalidomide) (Experimental): Patients receive pomalidomide PO QD on days 1-21. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After 12 cycles, patients with CR or PR continue pomalidomide for an additional 12 cycles with the option to continue thereafter in the absence of disease progression or unacceptable toxicity. After 12 cycles, patients with stable disease may continue pomalidomide for an additional 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray imaging throughout the trial. Patients may undergo CT as clinically indicated. Patients also undergo blood sample collection and may optionally undergo tissue biopsy during screening and on the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Pomalidomide; Procedure: X-Ray Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Pomalidomide — Given PO
  Other Names: 4-Aminothalidomide; Actimid; CC 4047; CC-4047; CC4047; Imnovid; Pomalyst
Procedure: X-Ray Imaging — Undergo x-ray imaging
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase II trial studies the effect of pomalidomide in treating patients with Kaposi sarcoma. Pomalidomide is a cancer fighting drug that stops the growth of blood vessels, stimulates the immune system, and may kill cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the proportion of participants with Kaposi sarcoma (KS) (with or without human immunodeficiency virus [HIV], regardless of previous treatment status) treated with pomalidomide who respond to treatment with a durable response (i.e., response duration of at least one year).

SECONDARY OBJECTIVES:

I. To measure the overall response rate (ORR) and report 95% confidence intervals in the overall study population.

Ia. To measure the ORR in the HIV positive study population. Ib. To measure the ORR in the HIV unrelated study population. II. To estimate the ORR in subgroups of KS in regard to HIV and previous treatment status.

III. To assess the safety of pomalidomide therapy. IV. To describe changes in visceral disease among those presenting with evaluable visceral disease.

EXPLORATORY OBJECTIVES:

I. To assess the effect of pomalidomide treatment on the tumor microenvironment and explore the relationship with clinical response.

II. To describe the effects of pomalidomide on CD4 lymphocyte counts and HIV viral load in HIV positive (+) participants.

III. To assess the effect of pomalidomide treatment on serum biomarkers and explore the relationship with clinical response.

IV. To assess Kaposi's sarcoma-associated herpesvirus (KSHV) viral copy number in plasma and explore whether changes correlate with clinical outcome.

OUTLINE:

Patients receive pomalidomide orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity. After 12 cycles, patients with complete response (CR) or partial response (PR) continue pomalidomide for an additional 12 cycles with the option to continue thereafter in the absence of disease progression or unacceptable toxicity. After 12 cycles, patients with stable disease may continue pomalidomide for an additional 12 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo chest x-ray imaging throughout the trial. Patients may undergo computed tomography (CT) as clinically indicated. Patients also undergo blood sample collection and may optionally undergo tissue biopsy during screening and on the trial.

After completion of study treatment, patients are followed up every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Participant is able to understand and willing to sign a written informed consent document
* Participants must have histologically or cytologically confirmed cutaneous KS. Participants must have measurable disease with a minimum of five bi-dimensionally measurable KS cutaneous marker lesions. If fewer than five bi-dimensionally measurable marker lesions are available, the total surface area of the marker lesion(s) must be >= 700 mm^2
* Participants must have documentation of HIV status

  * If HIV negative, documentation of a negative HIV rapid test within 21 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step).
  * If HIV positive, documentation of HIV-1 infection by means of any one of the following:

    * Documentation of HIV diagnosis in the medical record by a licensed health care provider
    * Documentation of receipt of antiretroviral therapy (ART) (at least two different medications that do not constitute a prescription for pre-exposure prophylaxis [PrEP]) by a licensed health care provider. Documentation may be a record of an ART prescription in the participant's medical record, a written prescription in the name of the participant for ART, or pill bottles for ART with a label showing the participant's name
    * Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multi-spot antibody differentiation assay
  * Note: The term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally (e.g., United States [U.S.] Food and Drug Administration [FDA])
  * WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an enzyme (E)/carbon immunoassay (CIA) that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 ribonucleic acid (RNA) viral load
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of pomalidomide in participants < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Life expectancy of greater than 6 months
* Hemoglobin >= 8 g/dL (within 14 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Absolute neutrophil count (ANC): >= 1,000/mm^3 (within 14 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Platelets: >= 75,000/mm^3 (within 14 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Bilirubin =< 1.5: x upper limit of normal (ULN) unless the patient is receiving an ART drug known to be associated with increased bilirubin, in which case the direct fraction should be =< 2 x ULN (within 14 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (within 14 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Serum creatinine =< 2.0 mg/dL/176.8 umol/L; or estimated creatinine clearance >= 15 mL/minute (1.00 mL/s) (as calculated per the Cockcroft-Gault equation (within 14 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Females of childbearing potential (FCBP), defined as a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally post menopausal for at least 24 consecutive months, i.e., has had menses at any time in the preceding 24 consecutive months) must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All patients must be counseled at a minimum of every 28 (± 2) days about pregnancy precautions and risks of fetal exposure
* HIV positive participants must be taking stable ART for >= 12 weeks, and have an undetectable HIV viral load within 28 days before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step). Minor fluctuations up to 200 copies/mL are acceptable
* HIV positive participants must not show recent improvement on ART that may confound response evaluation, within the following parameters:

  * If on ART 12 to 24 weeks, participants must show evidence of KS progression requiring further systemic treatment

    * Evidence of KS progression for eligibility include: Any new lesion(s); spreading of lesions by any measurable degree; development of ulceration; worsening edema documented by circumferential measure of limb or body; increase in symptoms such as pain, including negative psychological impact, requiring; any degree disease worsening by imagining) that would prompt expert assessment to recommend further systemic treatment without delay
  * If on ART for > 24 weeks, must show no evidence of regression in last 8 weeks

    * Evidence of KS regression for eligibility include: Measures of edema, lesion size or number, resolution of ulceration, or 20% improvement by imaging in largest diameter. For purposes of this assessment, if there is 20% reduction in size of any lesion, disappearance of any lesion, this constitutes regression unless there is concomitant increase in size or appearance of new lesions elsewhere
* Participants must agree to participate in and comply with the mandatory POMALYST Risk Evaluation and Mitigation Strategy (REMS) program
* Participants must be able to take aspirin 81 mg daily as prophylactic anticoagulation (patients intolerant to acetylsalicylic acid [ASA], may use one of the alternatives
* For participants with impaired decision-making capacity (IDMC): Participants with IDMC may be eligible for the study provided all other eligibility criteria are satisfied:

  * The participant's legally authorized representative (LAR) is able and willing to sign consent in addition to the study candidate
  * Both participant and LAR agree to follow study parameters and ensure that drug is taken per protocol, recorded in the study drug diary, and returned to clinic with any unused pills

Exclusion Criteria:

* Participant who is receiving any other investigational agents
* Participant has symptomatic visceral KS involving the lungs or gastrointestinal (GI) tract that requires immediate chemotherapy or radiotherapy. Participants with minimally symptomatic visceral disease not requiring immediate tumor shrinkage are eligible if in provider judgment potential disease progression will not cause a hazard for the participant
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pomalidomide
* Use of agents containing zidovudine (including Combivir and Trizivir) are prohibited. Changes to ART therapy during the study may be made if medically necessary (toxicity, failure of regimen, etc.). Use of medications or substances that are strong inhibitors of cytochrome P450 (CYP)1A2, which include amiodarone, cimetidine, fluoroquinolones (e.g., ciprofloxacin, enoxacin), fluvoxamine, and ticlopidine is prohibited. Co-administration of efavirenz, an inhibitor of CYP1A2, with strong inhibitors of CYP3A4 and P-glycoprotein (P-gp) is prohibited. Use of erythropoietin is prohibited. Co-administration of corticosteroids greater than doses required for treatment of adrenal insufficiency is prohibited. Because the lists of these agents are constantly changing, it is important to regularly consult frequently updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information. As part of the informed consent/enrollment procedures, the participant will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the participant is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection for which the participants have not completed at least 14 days of therapy prior to study enrollment into OPEN Step-1 (Treatment Assignment - Registration Step) and/or is not clinically stable
* Participant has symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
* Pregnant women are excluded from this study because pomalidomide is a thalidomide analog with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pomalidomide, breastfeeding should be discontinued if the mother is treated with pomalidomide
* Participants who have had chemotherapy, radiotherapy, or therapies to target KS lesions within 4 weeks (6 weeks for nitrosoureas or mitomycin C) with the exception of ART, before enrollment into OPEN Step-1 (Treatment Assignment - Registration Step)
* Participants with high clinical suspicion of concurrent Castleman disease or IL6 related inflammatory disease

  * For a reference of signs and symptoms consistent with IL6 related inflammatory disease or KSHV inflammatory cytokine syndrome (KICS) can refer to publication from Polizzotto Minnesota (MN), et al. Clinical Features and Outcomes of Patients with Symptomatic Kaposi Sarcoma Herpesvirus (KSHV)-associated Inflammation: Prospective Characterization of KICS. Clinical Infectious Diseases, 2016. 62(6):730-8
* Participants with a history of malignant tumors other than KS, unless:

  * In complete remission for >= 1 year, or
  * Completely resected basal cell or squamous skin carcinoma, or
  * In situ squamous cell carcinoma (SCC) of the cervix or anus
* Participants with grade >= 3 peripheral neuropathy
* Participants with a history of venous or arterial thromboembolism, unless line-rated thrombosis without embolus occurring >= 1 year prior to study entry
* Participants with a known procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein C deficiency, protein S deficiency, or antiphospholipid syndrome, but not including heterozygosity for the Factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome
* Participants with any prior use of pomalidomide, lenalidomide or thalidomide
* Participants with any condition, including the presence of laboratory abnormalities, which in the opinion of the responsible investigator places the participant at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Duration of response | From the first date at which a partial or complete response is documented until progression or death due to any cause, assessed up to 5 years
  The Kaplan-Meier (K-M) method will be used to describe duration of response for all treated participants. The cumulative proportion of study participants still in response at one year will be estimated using the point estimate and the 95% confidence interval using Greenwood's formula for the standard error of the K-M estimate. The proportional hazards model will be used to evaluate the association of human immunodeficiency virus (HIV) status and pretreatment status on duration of response.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 5 years post treatment
  The binomial proportion and its 95% confidence interval will be used to estimate ORR in four groups defined by HIV status and pretreatment status (HIV+, pretreated; HIV+, treatment naive; HIV-, pretreated and HIV-, treatment naive). In addition, the binomial proportion and its 95% confidence interval will be used to describe the ORR for HIV+ and HIV- participants, and those that were pretreated and treatment naïve.
Incidence of adverse events | Up to 5 years post treatment
  Will be assessed using version Common Terminology Criteria for Adverse Events 5.0. Adverse events observed on this study will be summarized by organ system, severity grade and relationship to pomalidomide. Frequency and severity of adverse events will be tabulated at the event and person level.
Changes in visceral disease | Baseline up to 5 years post treatment
  For those with evaluable visceral disease, changes in visceral disease will be descriptively reported.
Response duration in participants treated with pomalidomide | From the first date of which a partial or complete response is documented until first date of progression, assessed up to 5 years
  For deaths unrelated to progressive disease, duration of response will be censored at the date of the last Kaposi sarcoma (KS) evaluation during which the participant was determined to still be in response.

OTHER OUTCOMES:
Effect of treatment on changes in tumor microenvironment | Baseline up to 5 years post treatment
  Will assess the effect of pomalidomide treatment on the tumor microenvironment and explore the relationship with clinical response and summarize over time. Descriptive statistics for changes in tumor micro-environment will be calculated for all participants and according to clinical response to examine pre- and post-treatment differences and to explore the relationship with clinical response. Changes from baseline will be explored with one-sample nonparametric tests.
Effect of pomalidomide on CD4 lymphocyte counts | Up to within 7 days of treatment discontinuation
  Will be summarized over time.
Effect of pomalidomide on HIV viral load | Up to within 7 days of treatment discontinuation
  Will be summarized over time.
Change in Kaposi's sarcoma-associated herpesvirus (KSHV) viral copy number | Baseline up to within 7 days of treatment discontinuation
  Will assess KSHV viral copy number in plasma and explore whether changes correlate with clinical outcome and summarize this data over time. Descriptive statistics for changes in KSHV viral copy number will be calculated for all patients and according to clinical response to examine pre- and post-treatment differences and to explore the relationship with clinical response. Changes from baseline will be explored with one-sample nonparametric tests
Effect of pomalidomide on change in serum biomarkers | Baseline up to within 7 days of treatment discontinuation
  Will assess the effect of pomalidomide treatment on serum biomarkers and explore the relationship with clinical response and summarize this data over time. Descriptive statistics for changes in serum biomarkers will be calculated for all patients and according to clinical response to examine pre- and post-treatment differences and to explore the relationship with clinical response. Changes from baseline will be explored with one-sample nonparametric tests.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha L Vogt, Principal Investigator — AIDS Malignancy Consortium
Locations (15):
- United States (15):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Miami Cancer Institute, Miami, Florida
  - University of Illinois, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Mount Sinai Hospital, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Street at Quentin Mease Health Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Virginia Mason Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm